CLINICAL TRIAL: NCT05384158
Title: Evaluating Overlap and Distinctiveness in Neurocomputational Loss and Reward Elements of the RDoC Matrix
Brief Title: Valuation in Depressed Mood, Anhedonia, and Anxiety
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Virginia Polytechnic Institute and State University (Other)
Responsible Party: Principal Investigator, Pearl Chiu, Professor, Virginia Polytechnic Institute and State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: RDOC
Record Dates: First submitted 2022-05-13; First posted 2022-05-20 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-09

CONDITIONS: Neurobehavioral Components of Reward and Loss Valuation
Keywords: depression; anxiety; anhedonia
MeSH Terms: conditions — Depression; Anxiety Disorders; Anhedonia | interventions — Cognitive Behavioral Therapy; Educational Status

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Cognitive behavioral therapy (Active Comparator): cognitive behavioral therapy for depression, anxiety, and/or anhedonia
  Interventions: Behavioral: cognitive behavioral therapy
- Valuation with instruction (Active Comparator): repeat laboratory sessions of a reward/loss learning computer game with specific instructions
  Interventions: Behavioral: valuation with instruction
- Valuation without instruction (Active Comparator): repeat laboratory sessions of a reward/loss learning computer game without specific instructions
  Interventions: Behavioral: valuation without instruction

INTERVENTIONS:
Behavioral: cognitive behavioral therapy — cognitive behavioral therapy
  Arms: Cognitive behavioral therapy
Behavioral: valuation with instruction — repeat laboratory sessions of computerized learning game
  Arms: Valuation with instruction
Behavioral: valuation without instruction — repeat laboratory sessions of computerized learning game
  Arms: Valuation without instruction

SUMMARY:
This study examines how people respond to rewards and losses, and the extent to which these responses are linked or distinct among people experiencing depressed mood, anhedonia, and/or anxiety.

DETAILED DESCRIPTION:
This study tests relationships among neural and behavioral valuation mechanisms, and how these mechanisms change (or not) over time, with task instructions, and following cognitive behavior therapy.

ELIGIBILITY:
Inclusion Criteria:

* mood, anxiety, or anhedonia symptoms that affect functioning; fluent in English; able to see computer display; able to perform simple computer games.

Exclusion Criteria:

* history of seizure disorder, stroke, or head injury with more than 10 minutes of unconsciousness; hormone disorder; electroconvulsive therapy within 5 years; history of chemotherapy for cancer; current pregnancy; contraindications to MRI

Ages: 25 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 252 (Estimated)
Dates: Start 2021-08-01 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
change in proportion correct on the 'N-arm bandit learning task' | study entrance to study exit, an average of 12 weeks
  change in proportion correct on 'N-arm bandit reinforcement learning task' from study entrance to study exit

SECONDARY OUTCOMES:
change in depression symptoms (Beck Depression Inventory) | study entrance to exit, an average of 12 weeks
  change in depression symptoms from study entrance to study exit
change in anxiety symptoms (anxiety subscale; Mood and Anxiety Symptom Questionnaire) | study entrance to exit, an average of 12 weeks
  change in anxiety symptoms from study entrance to study exit
change in anhedonia symptoms (anhedonia subscale; Mood and Anxiety Symptom Questionnaire) | study entrance to exit, an average of 12 weeks
  change in anhedonia symptoms from study entrance to study exit

CONTACTS AND LOCATIONS:
Locations (1):
- Fralin Biomedical Research Institute at Virginia Tech Carilion, Roanoke, Virginia, United States

IPD SHARING:
Plan to Share IPD: No